CLINICAL TRIAL: NCT02357420
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of RM-131 Administered to Patients With Vomiting Symptoms and Moderate to Severe Diabetic Gastroparesis
Brief Title: Safety and Efficacy of Relamorelin Administered to Participants With Vomiting Symptoms and Moderate to Severe Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM-131-009; 2014-005623-27 (EudraCT Number)
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus Complications; Gastroparesis
Keywords: Diabetes Mellitus; Delayed Gastric Emptying; Vomiting; Gastroparesis; Gastrointestinal Motility Disorder
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications; Gastroparesis; Vomiting | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Relamorelin 10 μg (Experimental): Relamorelin 10 microgram (μg) was administered subcutaneously (SC) by injection twice daily (BID) for 12 weeks.
  Interventions: Drug: Relamorelin
- Relamorelin 30 μg (Experimental): Relamorelin 30 μg was administered SC by injection BID for 12 weeks.
  Interventions: Drug: Relamorelin
- Relamorelin 100 μg (Experimental): Relamorelin 100 μg was administered SC by injection BID for 12 weeks.
  Interventions: Drug: Relamorelin
- Placebo (Placebo Comparator): Placebo-matching relamorelin was administered SC by injection BID for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Relamorelin — Double blind relamorelin was given subcutaneously BID for 12 weeks.
  Other Names: RM-131
  Arms: Relamorelin 10 μg; Relamorelin 100 μg; Relamorelin 30 μg
Drug: Placebo — Placebo given subcutaneously for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of multiple dose regimens of relamorelin on vomiting episodes, gastric emptying and gastroparesis symptoms in participants with Type 1 and Type 2 diabetes mellitus and gastroparesis. Study drug (relamorelin and placebo) will be administered subcutaneously in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (T1DM) or Type 2 diabetes mellitus (T2DM) with stable glycemic control and Hemoglobin A1c (HbA1c) ≤11% at screening.
* Diabetic gastroparesis (DG), defined as at least a 3-month history of symptoms suggestive of gastroparesis on an ongoing basis (e.g., vomiting, nausea, early satiety, bloating, or epigastric or abdominal pain).
* Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD) score ≥2.6 at least once during the Screening Period (Visits 1-2).
* At least 2 vomiting episodes during the ~2 weeks prior to the first screening visit (Visit 1), as ascertained by patient history.
* Delayed Gastric Emptying (GE) confirmed at screening by abnormal Gastric Emptying Breath Test (GEBT), defined as GE half-time (t1/2) ≥79 minutes (the 80th percentile of normative data). At least 50% of patients enrolled will have a t1/2 ≥97 minutes (i.e., the 95th percentile).
* Stable concomitant medications, defined as no changes in regimen for at least 2 weeks prior to Visit 2 (daily adjustments of insulin doses are permitted).
* No use of metoclopramide, erythromycin, domperidone, or other gastrointestinal (GI) motility agents, or anti-emetics for at least 2 weeks prior to Visit 2, and willingness to remain off these medications (except as used as part of protocol-specific rescue medication) during the course of the clinical trial.
* Body mass index >18 kg/m2.
* If female, has a negative serum or urine pregnancy test and is not lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. Female patients unable to bear children must have this documented in the electronic case report form (eCRF) (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of 1 year since the last menstrual period]). Post-menopausal status will be confirmed by measurement of follicle stimulating hormone (FSH).
* Able to provide written informed consent prior to any study procedures and willing and able to comply with study procedures.

Additional inclusion criteria for randomization after the 2-week single-blind placebo run-in period:

* Compliance with the completion of the Diabetic Gastroparesis Symptom Severity Diary (DGSSD) and study drug injections, defined as approximately 80% diary completions and approximately 80% administration of injections, during the 2-week single-blind placebo run-in period. For those patients whose compliance is measured to be <80%, the final decision to randomize a patient will be made by the Investigator and the Sponsor (or designee).
* At least one vomiting episode at any time during the 2-week single-blind placebo run-in period, as recorded in the DGSSD.

Exclusion Criteria:

* Currently receiving parenteral feeding or presence of a nasogastric or other enteral tube [e.g., Percutaneous Endoscopic Gastrostomy (PEG) tube] for feeding or decompression.
* History of gastric surgery such as fundoplication, gastrectomy, gastric pacemaker placement, vagotomy, or bariatric procedure. (A history of diagnostic endoscopy is not exclusionary.)
* History of pyloric injection of botulinum toxin within 6 months of screening.
* Patients with clinical suspicion of upper GI obstruction (e.g., peptic stricture) must have been evaluated per standard of care and obstruction ruled out before screening.
* Currently taking opiates, or expecting to use opiates during the course of the clinical trial.
* Currently taking Glucagon-like peptide-1 (GLP-1) agonists, Sodium-glucose co-transporter 2 (SGLT2) inhibitors or pramlintide.
* Allergic or intolerant of egg, wheat, milk, or algae, as these are components of the Gastric emptying breath test (GEBT) study meal. (Gluten-free crackers can be provided.)
* History of anorexia nervosa, binge-eating, or bulimia within 5 years of screening.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN) at Visit 1.
* History of intestinal malabsorption or pancreatic exocrine disease.
* Requires hemodialysis or has end-stage renal disease.
* History of human immunodeficiency virus (HIV) infection.
* Clinically significant neurologic or psychiatric disorders that are likely to impact compliance with protocol requirements.
* Poor venous access or inability to tolerate venipuncture.
* Participation in a clinical study within the 30 days prior to dosing in the present study.
* Any other reason that, in the Investigator's opinion, would confound proper interpretation of the study or expose a patient to unacceptable risk, including renal, hepatic or cardiopulmonary disease, or significant acute electrocardiogram (ECG) abnormalities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2016-06-09 (Actual); Study Completion 2016-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wieslaw Bochenek, MD, Study Director — Allergan
Locations (98):
- United States (70):
  - Digestive Health Specialist of the Southeast, Dothan, Alabama
  - Huntsville, Alabama
  - Desert Sun Clinical Research, Tucson, Arizona
  - Adobe Clinical Research, Tucson, Arizona
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - Arkansas Primary Care Clinic, Little Rock, Arkansas
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - TriWest Research Associates, El Cajon, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Axis Clinical Trials, Los Angeles, California
  - Inland Empire Liver Foundation, Rialto, California
  - Syrentis Clinical Research, Santa Ana, California
  - Ventura Clinical Trials, Ventura, California
  - Danbury Hospital- Office of Clinical trials, Danbury, Connecticut
  - Avail Clinical Research, DeLand, Florida
  - International Research Associates LLC, Hialeah, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - APF Research, LLC, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Baptist Diabetes Associates, P.A., Miami, Florida
  - Miami, Florida
  - International Research Associates LLC, Miami, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - River Birch Research Alliance LLC, Blue Ridge, Georgia
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Medisphere Medical Research Center, Evansville, Indiana
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - Delta Research Partners, Monroe, Louisiana
  - Clinical Trials of America LA, LLC, West Monroe, Louisiana
  - Metropolitan Gastroenterology Group, P.C. (Chevy Chase Clinical Research) Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Detroit Clinical Research Center, PC-Farmington Hills, Farmington Hills, Michigan
  - Center For Digestive Health, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Planters Clinic, Port Gibson, Mississippi
  - Impact Clinical Trials, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Great Neck, New York
  - New York Clinical Trials, Inc, New York, New York
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - OnSite Clinical Solutions- Lexington OnSite Clinical Solutions, LLC, Lexington, North Carolina
  - Diabetes and Endocrinology Consultants, P.C., Morehead City, North Carolina
  - OnSite Clinical Solutions, LLC, Statesville, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Wake Forest University Baptist Health - Dept of Gastroenterology Medical Center Blvd, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - MetroHealth Medical Center, Leveland, Ohio
  - Great Lakes Gastroenterology Research, Mentor, Ohio
  - Northwest Gastroenterology Clinic, Portland, Oregon
  - Family Medicine of SayeBrook, Myrtle Beach, South Carolina
  - ClinSearch LLC, Chattanooga, Tennessee
  - El Paso, Texas
  - GI Specialists of Houston, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center & Medical School at Houston, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Gulf Coast Medical Research, LLC, Sugar Land, Texas
  - Aspen Clinical Research, Orem, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Khan and Abbasi Research, Chester, Virginia
  - Healing Hands of Virginia LLC, Richmond, Virginia
  - Gastroenterology Consultants, Virginia Beach, Virginia
  - ZainResearch, LLC, Richland, Washington
- Belgium (2):
  - Hopital Erasme - Universite Libre de Bruxelles, Brussels
  - UZ Leuven, Leuven
- Germany (5):
  - Herz und Diabeteszentrum Nordrhein Westfalen, Universitätsklinikum der Ruhr-Universiät Bochum, Bad Oeynhausen
  - Praxis Dr. Ott Rabenauer Str., Dippoldiswalde
  - GWT-TUD GmbH, Dresden
  - Israelitisches Krankenhaus Orchideenstig, Hamburg
  - Diabetes Zentrum und Praxis Prof. Pfützner Parcusstr., Mainz
- Israel (4):
  - Rambam Health Care Campus - Inst. of Endocrinology, Diabetes, and Metabolism, Haifa
  - Wolfson Medical Center, Holon
  - Rabin Medical Center, Beilinson Hospital Gastroenterology Dept, Petah Tikva
  - ZIV Medical Center, Safed
- Poland (8):
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Osteoporozy i Chorób Kostno-Stawowych J. Badurski S.J. ul., Bialystok
  - NZOZ Witamed al., Kielce
  - CenterMed Krakow, Krakow
  - Gabinet Lekarski dr n.med. Malgorzata Saryusz-Wolska ul., Lodz
  - NZOZ Pulsmedica ul., Lodz
  - KO-MED Centra Kliniczne, Staszów
  - Centrum Badawcze Wspólczesnej Terapii ul., Warsaw
  - Warsaw
- Sweden (2):
  - Gastroenterology Karolinska University Hospital Karolinska Universitetssjukhuset Gastro Centrum Medicine, Stockholm
  - Uppsala University Hospital Gastroenterology / Mag-Tarmmottagningen ingang, Uppsala
- United Kingdom (7):
  - NHS Tayside, Dundee, Scotland
  - Wansbeck General Hospital (Northumbria NHS Trust), Ashington
  - University Hospital of North Durham University Hospital of North Durham Research and Development Directorate, Durham
  - Royal Liverpool University Hospital, Liverpool
  - King's College Hospital, London
  - The James Cook University Hospital, Middlesbrough
  - Tyne and Wear

REFERENCES:
- [Derived] Camilleri M, Lembo A, McCallum R, Tourkodimitris S, Kemps L, Miller MB, Bertelsen K, Iacob A. Overall safety of relamorelin in adults with diabetic gastroparesis: Analysis of phase 2a and 2b trial data. Aliment Pharmacol Ther. 2020 Jun;51(11):1139-1148. doi: 10.1111/apt.15711. Epub 2020 Apr 17. PMID 32301137
- [Derived] Camilleri M, McCallum RW, Tack J, Spence SC, Gottesdiener K, Fiedorek FT. Efficacy and Safety of Relamorelin in Diabetics With Symptoms of Gastroparesis: A Randomized, Placebo-Controlled Study. Gastroenterology. 2017 Nov;153(5):1240-1250.e2. doi: 10.1053/j.gastro.2017.07.035. Epub 2017 Jul 29. PMID 28760384

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 393 participants were randomized and received study treatment, and 334 participants completed the study. Five participants who received study drug but discontinued prematurely were summarized as completing the study because they fulfilled the Visit 8 (Week 12) assessments as per protocol.
Groups:
- Placebo: Placebo-matching relamorelin was administered subcutaneously (SC) by injection twice daily (BID) for 12 weeks.
- Relamorelin 10 μg: Relamorelin 10 microgram (μg) was administered SC by injection BID for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Relamorelin 10 μg | Relamorelin 30 μg | Relamorelin 100 μg
Started | 104 | 98 | 109 | 82
Full Analysis Set (FAS) | 104 | 98 | 109 | 81 (1 participant from safety set did not enter FAS.)
Completed | 92 (3 participants who discontinued prematurely were included in completed as they fulfilled Visit 8.) | 86 (1 participant who discontinued prematurely was included in completed as he/she fulfilled Visit 8.) | 93 (1 participant who discontinued prematurely was included in completed as he/she fulfilled Visit 8.) | 63
Not Completed | 12 | 12 | 16 | 19
Not completed — Adverse Event | 3 | 3 | 8 | 9
Not completed — Investigator Decision | 1 | 0 | 0 | 0
Not completed — Prohibited Medication | 1 | 1 | 0 | 0
Not completed — Protocol Non-compliance | 0 | 0 | 0 | 1
Not completed — Withdrawn Consent | 4 | 8 | 6 | 6
Not completed — Lost to Follow-up | 3 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Safety Set (SS) included all participants who were randomized and received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Relamorelin 10 μg | Relamorelin 30 μg | Relamorelin 100 μg | Total
Number analyzed (Participants) | 104 | 98 | 109 | 82 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.9) | 59.3 (10.2) | 56.0 (11.7) | 57.1 (11.0) | 57.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 59 | 65 | 57 | 245
  Male | 40 | 39 | 44 | 25 | 148

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Weekly Vomiting Episodes
Description: Vomiting episodes were assessed via the Diabetic Gastroparesis Symptoms Severity Diary (DGSSD). The DGSSD is a 7-item, participant-reported daily diary designed to assess the severity of 6 core signs and symptoms of Diabetic Gastroparesis (DG) (nausea, abdominal pain, postprandial fullness, bloating, vomiting, and early satiety) and the frequency of vomiting episodes. Each day, the participant recorded the number of vomiting episodes in the past 24 hours in the diary. Higher scores indicate more vomiting episodes. Weekly scores were averaged across the 12 weeks period. A negative change from Baseline indicates improvement.
Time Frame: 7 days prior to Day 1 for Baseline to 7 days prior to Week 12
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study treatment and provided at least 1 postbaseline primary efficacy measurement (DGSSD). Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: vomiting episodes per week
Arm/Group | Placebo | Relamorelin 10 μg | Relamorelin 30 μg | Relamorelin 100 μg
Number analyzed (Participants) | 104 | 98 | 109 | 81
vomiting episodes per week
  Baseline: number analyzed (Participants) | 85 | 81 | 86 | 56
  Baseline | 5.7 (6.0) | 7.7 (17.2) | 6.9 (10.3) | 4.8 (5.2)
  Change from Baseline to Week 12: number analyzed (Participants) | 85 | 81 | 86 | 56
  Change from Baseline to Week 12 | -2.9 (5.8) | -3.7 (12.5) | -3.8 (7.6) | -1.1 (13.5)
Statistical Analysis 1: Comparison: Placebo vs Relamorelin 10 μg; Test type: Superiority; p = 0.36, Measures mixed effects model (MMRM); MMRM analysis used treatment, week, treatment-by-week interaction as fixed factors and baseline values as the covariates
Statistical Analysis 2: Comparison: Placebo vs Relamorelin 30 μg; Test type: Superiority; p = 0.25, MMRM; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Relamorelin 100 μg; Test type: Superiority; p = 0.59, MMRM; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline to Week 12 in Weekly DGSSD 4-symptom Composite Score (Nausea, Bloating, Early Satiety, Abdominal Pain)
Description: The DGSSD is a 7-item, participant-reported daily diary designed to assess the severity of 6 core signs and symptoms of DG (nausea, abdominal pain, postprandial fullness, bloating, vomiting, and early satiety) and the frequency of vomiting episodes. Severity of nausea, bloating and abdominal pain, were assessed on a numerical rating scale of 0 to 10, with 0 equating to "no" (symptom) and 10 equating to "worst possible" (symptom). Early satiety was assessed on a 5-item scale with 1 being "Only 1 or 2 bites" and 5 being "All of a normal-sized meal"; symptom severity scores for this item were reversed and normalized to a range 0 to 10 for the development of the DGSSD 4-symptom Composite Score. The DGSSD 4-symptom Composite Score (Nausea, Bloating, Early Satiety, Abdominal pain) range is 0 to 40. Higher scores indicate worse condition. Weekly scores were averaged across 12 weeks period. A negative change from Baseline indicates improvement.
Time Frame: 7 days prior to Day 1 for Baseline to 7 days prior to Week 12
Population: FAS included all randomized participants who received at least 1 dose of study treatment and provided at least 1 postbaseline primary efficacy measurement (DGSSD). Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Relamorelin 10 μg | Relamorelin 30 μg | Relamorelin 100 μg
Number analyzed (Participants) | 104 | 98 | 109 | 81
score on a scale
  Baseline: number analyzed (Participants) | 88 | 86 | 91 | 63
  Baseline | 21.4 (6.7) | 21.8 (6.9) | 21.1 (6.0) | 22.3 (6.2)
  Change from Baseline to Week 12: number analyzed (Participants) | 88 | 86 | 91 | 63
  Change from Baseline to Week 12 | -5.4 (8.1) | -7.7 (7.8) | -7.5 (7.4) | -8.9 (8.3)

3. Secondary Outcome: Change From Baseline to Week 12 for Gastric Emptying (GE) as Measured by the Gastric Emptying Breath Test (GEBT) Half-time
Description: GE was measured via the GEBT and was reported as a time to half (t1/2) of the theoretical total GE. GEBT is a non-radioactive stable isotope breath test intended for measurement of GE of solids in participants. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Relamorelin 10 μg | Relamorelin 30 μg | Relamorelin 100 μg
Number analyzed (Participants) | 104 | 98 | 109 | 81
minutes
  Baseline: number analyzed (Participants) | 89 | 83 | 92 | 63
  Baseline | 127.1 (36.5) | 126.8 (37.6) | 128.6 (35.9) | 133.6 (35.4)
  Change from Baseline to Week 12: number analyzed (Participants) | 88 | 82 | 92 | 61
  Change from Baseline to Week 12 | 0.0 (38.5) | -12.7 (38.1) | -12.8 (36.5) | -13.6 (40.5)

ADVERSE EVENTS:
Time Frame: Up to 98 days
Description: Safety set included all the participants who were randomized and received at least 1 dose of study treatment.
Arm/Group | Placebo | Relamorelin 10 μg | Relamorelin 30 μg | Relamorelin 100 μg
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/98 | 0/109 | 1/82
Serious Adverse Events (participants affected / at risk) | 8/104 | 7/98 | 10/109 | 6/82
Other Adverse Events (participants affected / at risk) | 13/104 | 21/98 | 30/109 | 28/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | Relamorelin 10 μg (N=98) | Relamorelin 30 μg (N=109) | Relamorelin 100 μg (N=82)
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Median nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Traumatic hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | Relamorelin 10 μg (N=98) | Relamorelin 30 μg (N=109) | Relamorelin 100 μg (N=82)
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 7 | 6
Urinary tract infection (Infections and infestations) | 7 | 7 | 8 | 6
Blood glucose increased (Investigations) | 1 | 3 | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 5 | 10 | 10
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 5
Headache (Nervous system disorders) | 3 | 4 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.